CLINICAL TRIAL: NCT02026739
Title: The Impact of Different Intraoperative Supplemental Oxygen Administration on the Pulmonary Function Following Minimally Invasive Esophagectomy: A Prospective Randomized Controlled Clinical Trial
Brief Title: The Optimal Intraoperative Supplemental Oxygen Administration During Minimally Invasive Esophagectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan, Lijie (Other)
Responsible Party: Sponsor-Investigator, Tan, Lijie, Professor of Surgery; Vice Chief, Division of Thoracic Surgery, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ZSHTA2013001
Record Dates: First submitted 2013-10-31; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Oxygenation Index
Keywords: minimally invasive esophagectomy; pulmonary function
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- low supplemental oxygen concentration (Experimental): The group in which low supplemental oxygen concentration of 40% will be performed during minimally invasive esophagectomy.
  Interventions: Procedure: low supplemental oxygen concentration
- high supplemental oxygen concentration (conventional) (Active Comparator): The group in which high supplemental oxygen concentration (onventional) of 80% will be performed during minimally invasive esophagectomy.
  Interventions: Procedure: high supplemental oxygen concentration (conventional)

INTERVENTIONS:
Procedure: low supplemental oxygen concentration — low supplemental oxygen concentration would be used during the surgery
  Arms: low supplemental oxygen concentration
Procedure: high supplemental oxygen concentration (conventional) — high supplemental oxygen concentration would be used during the surgery
  Arms: high supplemental oxygen concentration (conventional)

SUMMARY:
The study hypothesized that a relative low oxygen concentration (40%) supplemental would be advantageous to protect the pulmonary function of patients, comparied with conventional high oxygen concentration (80%). Therefore we raise this prospective randomized controlled research.

DETAILED DESCRIPTION:
Patients underwent minimally invasive esophagectomy in Zhongshan Hospital of Fudan University will be enrolled and be randomizedly assigned to low oxygen concentration (40%) supplemental or high oxygen concentration(80%) supplemental group. Intra-operative and post-operative pressure of Oxygen in Arterial Blood will be examined, and the surgical outcome will be recorded in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Staged T1-3N0M0 esophageal cancer patients or: patients who were restaged as T1-3N0M0 esophageal cancer after neo-adjuvant therapy.
2. Patients underwent minimally invasive esophagectomy(Thoracolaparoscopic McKeown procedure).

Exclusion Criteria:

1. Patients with previous thoracic surgery history.
2. Patients with severe Co-morbidity.
3. Pulmonary function is abnormal in the examination before surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
The change of oxygenation index | Change from Baseline at post-operative Day1
  The change of oxygenation index is an important index to indicate the pulmonary function of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lijie Tan, MD, Study Director — Fudan University
Locations (1):
- Division of Thoracic Surgery & Anesthesiology, Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China